CLINICAL TRIAL: NCT07295028
Title: A Phase 1 Randomized, Placebo- and Comparator-controlled (Bivalent and Monovalent Components), Observer-blind Study in Older Adults to Evaluate the Safety, Reactogenicity, and Immunogenicity of 3 Dose-levels of VXB-251 (Trivalent), for the Prevention of LRTD Caused RSV, hMPV, PIV3 and to Assess Immunological Interference and Cross-reactivity.
Brief Title: Study of an RSV-hMPV-PIV3 Trivalent Vaccine Candidate VXB-251 in Older Adults
Acronym: VXB251-001
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Vicebio Australia Proprietary Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: VXB251-001
Record Dates: First submitted 2025-11-24; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-11

CONDITIONS: Lower Respiratory Tract Disease; Healthy Participants
Keywords: RSV; hMPV; PIV3; Multipathogen respiratory virus vaccines
MeSH Terms: interventions — Biological Products

STUDY DESIGN:
Intervention Model Description: Stage 1 is a sequential assignment followed by Stage 2 parallel assignment.
Who Masked: Participant, Investigator
Masking Description: Double
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- VXB-251, low dose (Experimental)
  Interventions: Biological: trivalent (RSV/hMPV/PIV3) vaccine candidate
- VXB-251, medium dose (Experimental)
  Interventions: Biological: trivalent (RSV/hMPV/PIV3) vaccine candidate
- VXB-251, high dose (Experimental)
  Interventions: Biological: trivalent (RSV/hMPV/PIV3) vaccine candidate
- VXB-241 (Experimental)
  Interventions: Biological: bivalent (RSV/hMPV) unlicensed comparator
- VXB-213 (Experimental)
  Interventions: Biological: monovalent (RSV) unlicensed comparator
- VXB-221 (Experimental)
  Interventions: Biological: Biological/Vaccine: monovalent (hMPV) unlicensed comparator
- VXB-232 (Experimental)
  Interventions: Biological: monovalent (PIV3) unlicensed comparator
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: trivalent (RSV/hMPV/PIV3) vaccine candidate — VXB-251 low dose, single, IM injection.
  Arms: VXB-251, low dose
Biological: trivalent (RSV/hMPV/PIV3) vaccine candidate — VXB-251 medium dose, single, IM injection.
  Arms: VXB-251, medium dose
Biological: trivalent (RSV/hMPV/PIV3) vaccine candidate — VXB-251 high dose, single, IM injection.
  Arms: VXB-251, high dose
Biological: bivalent (RSV/hMPV) unlicensed comparator — VXB-241 medium dose, single, IM injection.
  Arms: VXB-241
Biological: monovalent (RSV) unlicensed comparator — VXB-213 medium dose, single, IM injection.
  Arms: VXB-213
Biological: Biological/Vaccine: monovalent (hMPV) unlicensed comparator — VXB-221 medium dose, single, IM injection.
  Arms: VXB-221
Biological: monovalent (PIV3) unlicensed comparator — VXB-232 medium dose, single, IM injection.
  Arms: VXB-232
Other: Placebo — diluent, single, IM injection.
  Arms: Placebo

SUMMARY:
This study is being done to find out how safe and effective a new combined vaccine candidate, called VXB-251, is for older adults. The vaccine candidate is designed to protect against three common viruses that can cause respiratory tract infections:

* RSV (respiratory syncytial virus)
* hMPV (human metapneumovirus)
* PIV3 (parainfluenza virus type 3)

Two components of this vaccine (RSV and hMPV) have already been tested in people before, as part of another study for a two-in-one vaccine. However, this is the first time that the PIV3 component and all three components together (RSV, hMPV, and PIV3) are being tested in people.

The vaccine candidate will be given as a single intramuscular injection. The study will also test unlicensed comparator vaccines and a placebo (a substance that looks like the real vaccine but doesn't contain any active ingredients) that target none, one or two of these viruses to see whether combining all three components affects safety or how well the immune system responds.

DETAILED DESCRIPTION:
This is a multicenter randomized, placebo- and comparator-controlled, dose-ranging study to be conducted in Australia in older adults, aged 60 to 83 years, to evaluate the safety, reactogenicity, and immunogenicity of a trivalent RSV/hMPV/PIV3 vaccine candidate, VXB-251. All investigational medicinal products (IMPs) will be administered as a single 0.5 mL intramuscular injection on day 1.

Recruitment will be in 2 stages:

Stage 1 (N=10). Two cohorts, each of 5 participants, will be sequentially enrolled at a 4:1 ratio to receive:

* Cohort 1: either a medium dose of the vaccine candidate or the placebo control,
* Cohort 2: either a high dose of the vaccine candidate or the placebo control

At each enrolling site, at least 1 hour must elapse between IMP injection in the first sentinel and next IMP injection to monitor for hypersensitivity reactions and other fast-onset adverse events (AEs). The investigator or delegate will decide if and when the next sentinel can be vaccinated.

A Safety Monitoring Committee (SMC) will make recommendations on escalation from 1 sequential cohort to the next and progress from Stage 1 to Stage 2 based on 1-week safety and reactogenicity available data from the prior cohort.

Stage 2 (N=230). Participants will be concurrently assigned on day 1 (Visit 2) at an unequal ratio into 1 of 8 study groups and receive one of the following:

* VXB-251 trivalent (RSV/hMPV/PIV3) vaccine candidate, low dose (N=30)
* VXB-251 trivalent (RSV/hMPV/PIV3) vaccine candidate, medium dose (N=26)
* VXB-251 trivalent (RSV/hMPV/PIV3) vaccine candidate, high dose (N=26)
* VXB-241 bivalent (RSV/hMPV) unlicensed comparator (N=30)
* VXB-213 monovalent (RSV) unlicensed comparator (N=30)
* VXB-221 monovalent (hMPV) unlicensed comparator (N=30).
* VXB-232 monovalent (PIV3) unlicensed comparator (N=30)
* Placebo (N=28)

In Stage 1, the study will be open-label across cohorts and observer-blind within each cohort. In Stage 2, the study will be observer-blind.

The study duration for each participant will be 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 60 to 83 years of age at inclusion.
2. Evidence of signed and dated participant informed consent form (PICF) prior to any study procedure, indicating that the subject has been informed of all pertinent aspects of the study.
3. Willingness and ability to comply with the planned study visits and calls, procedures, and restrictions for the duration of the study.
4. Good health, which allows for pre-existing well controlled and low impact chronic diseases, except for the diseases listed in the exclusion criteria. A disease is defined as well controlled and has a low impact if it did not require meaningful change in therapy or unplanned medical visit(s) in the previous 3 months and allows participant's primary responsibility for self-care and daily living activities.
5. Non-smoker or occasional smoker, defined as smoking less than 10 nicotine-containing cigarettes/ vapes/cigars/pipe fills per week.
6. Contraception and childbearing/conception potential: only female participants with non-childbearing potential will be included. Male participants in a relationship with a female partner of childbearing potential must be willing to use a double contraceptive method together with their female partner for at least 4 weeks before and 12 weeks after the IMP injection at Visit 2 (day 1).
7. Body mass index (BMI) ≥ 17.0 kg/m2 and ≤ 35.0 kg/m2.

Exclusion Criteria:

1. History of RSV, hMPV, and/or PIV3 infection affecting the participant and/or the participant's household in the previous 12 months.
2. History of autoimmune disease (AID) or possibly autoimmune disease (pAID) requiring therapeutic intervention, even if stable and well controlled, including, but not limited to, systemic lupus erythematosus, autoimmune arthritis/rheumatoid arthritis, Guillain-Barré syndrome, multiple sclerosis, Sjögren's syndrome, idiopathic thrombocytopenia purpura, glomerulonephritis, autoimmune thyroiditis, temporal arteritis, psoriasis, insulin-dependent diabetes mellitus, celiac disease.
3. Confirmed or suspected immunodeficiency, even if stable and well controlled.
4. Ongoing severe asthma. Other allergic diseases (e.g., allergic rhinitis, atopic dermatitis / eczema, mild to moderate asthma, food allergies) are allowed at the investigator's or delegate's discretion.
5. History of significant allergic reaction (e.g., anaphylaxis, hypersensitivity, angioedema) to medication or food or known allergy to vaccine, or any excipients in the formulation, and latex.
6. History of severe AE associated with vaccine administration.
7. Ongoing disorders of coagulation, which contraindicate IM injections.
8. Donation or loss of ≥ 500 mL whole blood on the previous 2 months, and/or donation of plasma in the previous 1 week, and/or intention to donate blood or plasma during the study.
9. Positive serum test results indicating ongoing HIV, HBV and/or HCV infection, and/or documented ongoing HIV, HBV, or HCV infection.
10. Other poorly controlled and/or impactful chronic disease. A disease is defined as poorly controlled if it requires meaningful change in therapy and/or unplanned medical visit(s) in the previous 3 months. A disease is defined as impactful if, in the investigator's judgment, it meaningfully affects the participant's ability to manage self-care and/or activities of daily living.
11. Disease expected to prevent completion of the study (i.e. to rapidly deteriorate within the timeframe of the study).
12. Prior treatments.

    1. Receipt of licensed RSV vaccine and/or enrollment in clinical trials(s) evaluating investigational RSV, hMPV, PIV3, and/or molecular clamp-based vaccine candidates at any time, unless it was documented that the participant received a placebo.
    2. Other investigational drug or vaccine received in the previous 6 months.
    3. Chemotherapy, radiotherapy, and/or other immunosuppressive medication (including biologics) received in the previous 6 months.
    4. IgGs or any blood product received in the previous 3 months.
    5. Systemic corticosteroids (oral/intravenous/IM) at doses equivalent to ≥ 20 mg prednisone per day received for ≥ 14 days, even if not consecutive, during the previous 3 months. Inhaled/nebulized, intra-articular, intra-bursal, skin, and eye topical corticosteroids are permitted.
    6. Received or plan to receive licensed non-live vaccine(s) for the period starting 2 weeks before to 4 weeks after of the study IMP injection or licensed live vaccine(s) for the period starting from 4 weeks before to 4 weeks after the study IMP injection. Pandemic or emergency vaccines are always allowed as per country guidelines.
13. Clinically meaningful abnormal finding from physical examination, vital sign assessment, electrocardiogram (ECG), safety laboratory test results. If deemed appropriate, the investigator or delegate may repeat these assessments.
14. History of alcohol abuse in the previous year determined at the investigator's discretion.
15. History of recreational drug abuse in the previous year and/or positive test for drugs of abuse at Visit 2 (day 1), unless there is an explanation acceptable to the investigator (e.g., the participant has informed in advance that he/she consumed a prescription or over-the-counter product that contained the detected drug).
16. Intention to participate in any investigational drug/vaccine/medical device clinical trial at any time throughout the planned duration of this study.
17. Presence of tattoo, scarring, skin discoloration, or any other skin disturbances at the injection site which may interfere with effective assessment of the injection site.
18. Intention to move to a location that would prevent participating in the study until study end.
19. Any other reason which would prevent the participant from participating in the study or interfere with the participant's compliance with study procedures.

Ages: 60 Years to 83 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2026-05-24 (Estimated); Study Completion 2027-04-24 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants With 1 or More Unsolicited Adverse Events (AEs) | 1 month after IMP injection
Proportion of Participants With 1 or More Serious Adverse Events (SAEs), AEs of Special Interest (AESIs), and Premature Discontinuation Associated AEs (PDAEs) | 1 month after IMP injection
Proportion of Participants With 1 or More Solicited AEs | 7 days after IMP injection

SECONDARY OUTCOMES:
Proportion of Participants With Serious Adverse Events (SAEs), AEs of Special Interest (AESIs), and Premature Discontinuation Associated AEs (PDAEs) | 6 and 12 months after IMP injection
Proportion of Participants With 1 or More Severe Solicited AEs | 7 days after IMP injection
Geometric Mean Fold Increase (GMFI) of RSV-A, RSV-B, hMPV-A, hMPV-B, and PIV3 Serum Neutralizing Antibody Titers | Pre-injection baseline to 1 month, 6 months, and 12 months, after IMP injection
  GMFI is defined as geometric mean of ratios of specific antibody titer/concentration at each post-injection time point over pre-injection baseline.
Geometric Mean Titers (GMTs) of RSV-A, RSV-B, hMPV-A, hMPV-B, and PIV3 Serum Neutralizing Antibody Titers | Pre-injection baseline to 1 month, 6 months, and 12 months after IMP injection
Proportion of Participants with Sero-response Greater Than or Equal to (>=) 4-fold (SRR-4) and 8-fold (SRR-8) Increase from Baseline in Neutralizing Antibody Titers for RSV-A, RSV-B, hMPV-A, hMPV-B, and PIV3 | Pre-injection baseline up to 1 month, 6 months, and 12 months after IMP injection
GMFI of RSV PreF, hMPV PreF, and PIV3 PreF Serum Immunoglobulins G (IgG) Concentrations | Pre-injection baseline to 1 month, 6 months, and 12 months after IMP injection
Geometric Mean Concentrations (GMC) of RSV PreF, hMPV PreF, and PIV3 PreF Serum IgG | 1 month, 6 months, and 12 months after IMP injection
Geometric Mean Ratios (GMRs) of Fold Increase of RSV-A and RSV-B Neutralizing Serum Antibody Titers Versus Fold Increase of RSV PreF Serum IgG Concentration | Pre-injection baseline to 1 month, 6 months, and 12 months after IMP injection
GMR of Fold Increase of hMPV-A and hMPV-B Neutralizing Serum Antibody Titers Versus Fold Increase of hMPV PreF Serum IgG Concentration | Pre-injection baseline to 1 month, 6 months, and 12 months after IMP injection
GMR of Fold Increase of PIV3 Neutralizing Serum Antibody Titers Versus Fold Increase PIV3 PreF Serum IgG Concentration | Pre-injection baseline to 1 month, 6 months, and 12 months after IMP injection

CONTACTS AND LOCATIONS:
Overall Officials: Nischal Sahai, MD, Principal Investigator — University of the Sunshine Coast, South Bank; Stephanie Wallace, MD, Principal Investigator — University of the Sunshine Coast, Sippy Downs; Christopher Moller, MD, Principal Investigator — University of the Sunshine Coast, Morayfield; Rebecca Wolf, MD, Principal Investigator — Veritus Research; Madeleine Janin, MD, Principal Investigator — Momentum Clinical Research; Rishi Shah, MD, Principal Investigator — Emeritus Research
Locations (6):
- Australia (6):
  - University of Sunshine Coast, South Bank, Brisbane
  - Emeritus Research, Camberwell
  - Momentum Clinical Research, Darlinghurst
  - Veritus Research, Melbourne
  - University of the Sunshine Coast, Morayfield
  - University of the Sunshine Coast, Sippy Downs, Sippy Downs

IPD SHARING:
Plan to Share IPD: No